CLINICAL TRIAL: NCT02135822
Title: Phase II Trial of Nab-paclitaxel Plus Gemcitabine in First-line Treatment of Chinese Patients With Advanced Pancreatic Cancer
Brief Title: Nab-paclitaxel Plus Gemcitabine in Chinese Patients With Advanced Pancreatic Cancer
Acronym: NAPGAP
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Liu, Rong, Professor and chief physician, Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABX-LR001
Record Dates: First submitted 2014-05-08; First posted 2014-05-12 (Estimated); Last update posted 2014-05-16 (Estimated); Status verified 2014-05

CONDITIONS: Advanced Pancreatic Cancer
Keywords: nanoparticle albumin-bound paclitaxel; gemcitabine; advanced pancreatic cancer
MeSH Terms: interventions — Taxes; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- nanoparticle albumin-bound paclitaxel, gemcitabine (Experimental): Nanoparticle albumin-bound paclitaxel is given at 125 mg/m2 intravenously on day 1 and 8, in combination with gemcitabine which is given at 1000 mg/m2, on day 1 and 8, each 21-day cycle. Number of cycle: 6 cycles.
  Interventions: Drug: nanoparticle albumin-bound paclitaxel; Drug: gemcitabine

INTERVENTIONS:
Drug: nanoparticle albumin-bound paclitaxel — Nanoparticle albumin-bound paclitaxel is given at 120 mg/m2 intravenously on day 1 and 8 of each 21-day cycle. Number of cycles: 6 cycles.
  Other Names: nab-paclitaxel; Abraxane; ABI-007
Drug: gemcitabine — Gemcitabine is given intravenously at 1000 mg/m2 on day 1 and 8 of each 21-day cycle. Number of cycles: 6 cycles.
  Other Names: Gemzar

SUMMARY:
The purpose of this study is to determine the efficacy and safety of nanoparticle albumin-bound paclitaxel (nab-paclitaxel) plus gemcitabine as first-line treatment in Chinese patients with advanced pancreatic ductal adenocarcinoma.

DETAILED DESCRIPTION:
Advanced pancreatic ductal adenocarcinoma is a fatal disease with about 6 months of median overall survival (OS). Gemcitabine is the only approved single agent. Gemcitabine-based chemotherapy did not show benefit in OS during the past decade. The recent phase III trial MPACT (Metastatic Pancreatic Adenocarcinoma Clinical Trial) demonstrated an improvement in overall response rate (ORR), progression free survival (PFS) and OS, with nab-paclitaxel (125 mg/m2 on day 1, 8 and 15 every 28 days) plus gemcitabine (1000 mg/m2 on day 1, 8 and 15 every 28 days) compared to gemcitabine alone. Accordingly the combination of nab-paclitaxel with gemcitabine became one of standard treatments in metastatic pancreatic cancer. A Chinese phase II trial showed the modified dosage of nab-paclitaxel (120 mg/m2 on day 1 and 8 every 21 days) plus gemcitabine (1000 mg/m2 on day 1 and 8 every 21 days) is more suitable for Chinese patients. This study aims to explore the efficacy and safety of the tentative dosage of nab-paclitaxel (125 mg/m2 on day 1 and 8, every 21 days) and gemcitabine (1000 mg/m2 on day 1 and 8, every 21 days) for Chinese patients.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed-consent form.
2. Age no less than 18 years.
3. Histologically confirmed locally advanced or metastatic pancreatic ductal adenocarcinoma, with RECIST measurable lesions.
4. Eastern Cooperative Oncology Group (ECOG) 0-1 with life expectation of no less than 12 weeks.
5. Patients must have received no previous chemotherapy or investigational therapy for the treatment of metastatic disease. Prior treatment with 5-fluorouracil or gemcitabine administered as a radiation sensitizer in the adjuvant setting is allowed, provided at least 6 months have elapsed since completion of the last dose and no lingering toxicities are present.
6. Adequate liver/bone marrow function.
7. Human Chorionic Gonadotropin (HCG) test negative for female with contraception measure until 3 months after study end.
8. Compliant, and can be followed up regularly.

Exclusion Criteria:

1. Pregnant or breast-feeding female, or not willing to take contraception measures during study.
2. Serious infection requiring antibiotics intervention during recruitment.
3. Allergic to study drug.
4. More than grade 1 neuropathy.
5. Uncontrolled brain metastasis or mental illness.
6. Congestive heart failure, uncontrolled cardiac arrhythmia, etc.
7. Other malignancy within 5 years.
8. Can't be followed up or obey protocol.
9. Ineligible by the discretion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-05; Primary Completion 2015-05 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | Measure at every 6 weeks (every 2 cycles) up to 18 weeks
  Percentage of patients who achieve partial response (PR) or complete response (CR) based on Response Evaluation Criteria In Solid Tumors (RECIST).

SECONDARY OUTCOMES:
Progression-free survival | up to 15 months
  Measurement of time from study treatment to disease progression or death.
Overall survival | up to 2 years
  Measurement of time from study treatment to patient's death or lost to follow-up.
Disease control rate | Measure every 6 weeks (every 2 cycles) up to 18 weeks
  The sum of rates of partial response, complete response and steady disease based on Response Evaluation Criteria In Solid Tumors (RECIST).
Safety and tolerability | up to 18 month
  Percentage of patients who experience adverse events during this study.

CONTACTS AND LOCATIONS:
Overall Officials: Rong Liu, Principal Investigator — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Xu R, Yu X, Hao J, Wang L, Pan H, Han G, Xu J, Zhang Y, Yang S, Chen J, Ying J, Dai G, Li M, Begic D, Lu B, Shen L. Efficacy and safety of weekly nab-paclitaxel plus gemcitabine in Chinese patients with metastatic adenocarcinoma of the pancreas: a phase II study. BMC Cancer. 2017 Dec 22;17(1):885. doi: 10.1186/s12885-017-3887-z. PMID 29273007